CLINICAL TRIAL: NCT05630118
Title: Testing an Online Insomnia Intervention to Reduce Alcohol Use Via Improved Sleep Among Heavy Drinkers
Brief Title: Online Insomnia Intervention to Reduce Alcohol Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessica Weafer (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Jessica Weafer, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 60446-2; 1R21AA029201-01A1 (NIH)
Record Dates: First submitted 2022-11-17; First posted 2022-11-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Alcohol Use Disorder; Heavy Drinking
Keywords: Sleep; Cognitive Behavioral Therapy; CBT; Alcohol; App; Non Pharmacological
MeSH Terms: conditions — Alcoholism; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHUTi Intervention (Experimental): Adult heavy drinkers with insomnia
  Interventions: Behavioral: SHUTi Intervention
- Web-Based Insomnia Education Program (Active Comparator): Adult heavy drinkers with insomnia
  Interventions: Behavioral: Web-Based Insomnia Education Program

INTERVENTIONS:
Behavioral: SHUTi Intervention — Sleep Healthy Using the Internet (SHUTi) is a well-validated version of e-CBT-I comprised of 6 weekly educational modules and daily sleep diaries. Participants will have 9 weeks to complete 6 once-weekly educational "cores." Cores consist of: insomnia overview, sleep restriction, stimulus control, cognitive restructuring, sleep hygiene, and relapse prevention, and last approximately 45 minutes each. Participants will receive weekly objectives, as well as review and feedback on the previous core's assignments and sleep diary data, new material, assignments, and a summary. These features are supplemented with interactive features (i.e., personalized goal-setting, video vignettes). Participants receive daily emails prompting them to complete the 11-item sleep and alcohol use diary daily during the intervention.
  Arms: SHUTi Intervention
Behavioral: Web-Based Insomnia Education Program — Participants will be given access to a web-based program on sleep education to read at their own pace during the 9-week intervention period. The program content overlaps with SHUTi on the following topics: insomnia symptoms, impacts, and causes, basic sleep improvement strategies, and when to see a doctor. The information is akin to that found on WebMD or National Sleep Foundation website. Unlike the SHUTi program, the information is fixed, accessible immediately (no week-to-week information "unlocking") and there are no customized bedtime or wake-time suggestions based on sleep diary data.
  Arms: Web-Based Insomnia Education Program

SUMMARY:
Alcohol use disorder (AUD) inflicts enormous physical, emotional, and financial burdens on the individual and society at large. Insomnia is highly prevalent among individuals with AUD, and disrupted sleep contributes substantially to alcohol-related problems. While research suggests that treating insomnia may effectively reduce AUD, the degree to which treating insomnia in heavy drinkers reduces alcohol consumption and prevents the onset of severe AUD is not known. This study will be the first to evaluate an Internet-based version of cognitive behavioral therapy for insomnia (CBT-I) in community-dwelling, heavy drinking adults with insomnia. Sleep Healthy Using the Internet (SHUTi), the most widely-used and well-validated version of Internet-based CBT-I will be used. The primary aim is to reduce alcohol consumption and insomnia severity in this population.

DETAILED DESCRIPTION:
The study will investigate the efficacy of Sleep Healthy Using the Internet (SHUTi), an online insomnia intervention, in reducing alcohol consumption and improving sleep in heavy drinkers with insomnia. The participants are ages 18-50 (N=100) who have insomnia and are heavy drinkers (at least weekly binge drinking episodes [4/5+ drinks in one sitting for men/women]). This intervention has a mixed methods randomized controlled trial design. Participants will be randomly assigned to either the online SHUTi intervention (N=50), or a patient education (PE) website (N=50). Quantitative data will be collected via online REDCap surveys and daily online diaries. Qualitative data will be collected via semi-structured telephone interviews. Data collection points will be pre-intervention, post-intervention, and 3- and 6-months postintervention.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* Fluency in English
* At least weekly binge drinking episodes (4/5+ drinks for women/men)]
* Insomnia Severity Index (ISI) scores #15

Exclusion Criteria:

* No internet access
* Past or current substance use disorder (other than mild or moderate AUD)
* Obstructive sleep apnea
* Bipolar disorder, schizophrenia, or other psychotic spectrum disorder
* Pregnancy or nursing for women
* Any serious medical or neurological problems

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Change In Alcohol Use: Daily Alcohol Diaries | 33 weeks (baseline, at the end of the 9-week intervention, at 3- and 6-months post-intervention)
  Participants will report the number of drinks consumed each day and proximity of alcoholic drinks to bedtime. Summary measures will include total number of drinking days, total number of drinks, average number of drinks per drinking day, and total number of binge episodes (4/5+ drinks for women/men) over a 10-day period.
Change In Sleep: Insomnia Severity Index (ISI) | 33 weeks (baseline, at the end of the 9-week intervention, at 3- and 6-months post-intervention)
  The ISI uses a 7-item scale to asses insomnia impact over the previous two weeks. Items scores range from 0-28. Scores indicate moderate to severe insomnia. Moderate or marked clinical improvement is indicated by a change score of >7 or >8 respectively.
Change In Sleep: 2) Pittsburgh Sleep Quality Index (PSQI) | 33 weeks (baseline, at the end of the 9-week intervention, at 3- and 6-months post-intervention)
  The PSQI indexes one-month global sleep quality using 18 items scored on a scale from 0-21. Scores # 5 indicate poor sleep quality.
Change In Sleep: 3) Daily Sleep Diaries | 33 weeks (baseline, at the end of the 9-week intervention, at 3- and 6-months post-intervention)
  Sleep Onset Latency (SOL). Participants will report how long it took them to fall asleep.
Change In Sleep: 4) Daily Sleep Diaries | 33 weeks (baseline, at the end of the 9-week intervention, at 3- and 6-months post-intervention)
  Wake after Sleep Onset (WASO): Participants will report the number of minutes awake after falling asleep.
Change in Medication Use: 5) Daily Sleep Diaries | 33 weeks (baseline, at the end of the 9-week intervention, at 3- and 6-months post-intervention)
  Participants will report the amount of sleep medication used each day.

SECONDARY OUTCOMES:
Change In Mood: 1) Perceived Stress Scale (PSS) | 33 weeks (baseline, at the end of the 9-week intervention, at 3- and 6-months post-intervention)
  The PSS will assess perceived stress over the prior month. Scores range from 0-40. The PSS demonstrates strong concurrent and predictive validity for various health behaviors and outcomes with higher scores indicating greater psychological distress.
Change In Mood: 2) Center for Epidemiologic Studies Depression Scale-Revised (CESD-R-10) | 33 weeks (baseline, at the end of the 9-week intervention, at 3- and 6-months post-intervention)
  The CESD-R-10 will index past-week depressive symptoms. Scores range from 0-30. Higher scores represent more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Weafer, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University Of Kentucky Psychology Research Lab, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No